CLINICAL TRIAL: NCT05815147
Title: An Exploratory Real-world Study to Explore the Effects of Fortified Powdered Beverage on Sleep Quality in Chinese Adults with Mild Sleep Issue(s) or Complaint(s)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Nutricia (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NELN202209A
Record Dates: First submitted 2023-03-20; First posted 2023-04-18 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Sleep
Keywords: Mild Sleep Issue(s) or Complaint(s)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study Group (Experimental): Participants will be asked to take study product.
  Interventions: Dietary Supplement: Fortified Powdered Beverage

INTERVENTIONS:
Dietary Supplement: Fortified Powdered Beverage — Participants will be asked to take the fortified powdered beverage everyday for 6 weeks.

SUMMARY:
The goal of this exploratory study is to explore the sleep and related health benefits of the study product in Chinese middle-aged & elderly population in real world settings and potentially generate hypothesis on key exploratory and other exploratory objectives. The main questions it aims to answer are:

* To explore the effects of test product on sleep quality;
* To understand and evaluate effects of test product on sleep pattern;
* To assess the subjects' overall health status self-evaluation. etc.

Participants will be asked to take study product, collect the sleep pattern parameters and report the overall health status.

ELIGIBILITY:
Inclusion Criteria:

1. Adults older than 50 years of age;
2. Chinese ethnicity;
3. BMI is between 18 and 30 (excluding upper and lower bound values);
4. Mild sleep issue(s) and/or complaint(s), including but not limited to difficulty initiating sleep, difficulty maintaining sleep, increased number of nocturnal awakenings, early awakening, complaints of non-restorative sleep, dissatisfaction with sleep quality etc.;
5. PSQI score >7 at screening;
6. PHQ-4 score ≤ 3 at screening;
7. Sufficient ability in Chinese to complete informed consent and other study documents, and willingness to complete this study according to the study protocol;
8. Sufficient ability to install and use a secure WeChat platform on the mobile phone during the study period; stable connectivity to network through mobile phone;
9. Sufficient reading and writing and understanding ability in Chinese to complete questionnaires; daily diaries etc.;
10. Can be directly contacted by mobile phone or WeChat throughout the study;
11. Stable life status with no cross-provincial moving or job changing in the past 6 months, no intention to move or change job during study period.

Exclusion Criteria:

1. Currently receiving medication and other therapies for sleep disorders, including but not limited to sleeping pills and traditional Chinese medicine or therapies;
2. Predominant complaint(s) of parasomnia or sleep apnea and/or medically diagnosed primary sleep disorders including but not limited to obstructive sleep apnea (OSA), narcolepsy, periodic limb movement (PLMD), restless leg syndrome (RLS), or REM sleep behaviors disorder;
3. Long-term (≥3 months) use of drugs that induce sleep disturbances, including but not limited to CNS stimulants, anti-depressents, antipsychotics etc.;
4. Use sedative drugs within 4 weeks prior to screening;
5. Use of dietary supplements with sleep effects within 4 weeks prior to screening including but not limited to melatonin, GABA, Ziziphi Spinosa Semen etc.;
6. Average daily caffeinated drinks intake of 5 cups or more (200ml/cup) , including but not limited to coffee, tea, energy drinks, during 4 weeks prior to screening, or during the study period;
7. Allergic or intolerant to the ingredients of the investigational products, such as protein allergy, dairy allergy, lactose intolerance, soy allergy and fish allergy etc. ;
8. The presence of drug abuse or alcohol and/or psychoactive substances abuse;
9. Those who work night shifts or perform unusal working hours;
10. The presence of medical, psychological or social conditions that may interfere with the subject's participation in the study or affect the evaluation of the study results at the investigator's discretion;
11. Pregnant and lactating women, caregivers of newborns unsuitable for trial participation at the investigators' discretion;
12. Participation in any other studies involving investigational or marketed products concomitantly or two weeks prior to enrolment;
13. Do not agree to sign the informed consent.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-07-21 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
Sleep quality | 6 weeks
  Sleep quality is measured by Chinese version Pittsburgh Sleep Quality Score (CPSQI). The total score ranges from 0 to 21 points. The higher score indicates the worse sleep quality.

OTHER OUTCOMES:
total sleep time (TST) for Sleep pattern | 6 weeks
  Total sleep time, the amount of actual sleep time in a sleep episode; Unit: minute.
Number of wakening after sleep onset (WASO) for Sleep pattern | 6 weeks
  The number of wakening times during a sleep episode; Unit: time.
Heart Rate (HR) for Sleep pattern | 6 weeks
  Heart Rate (HR) during sleep episode; Unit: beats per minute (BPM).
Quality of life for overall health status self-evaluation | 6 weeks
  Quality of life Questionnaire: The World Health Organization Quality of Life - BREF (WHOQOL-BREF, Chinese version).
  WHOQOL - BREF scale includes 24 items of physical, psychological, social, and environmental in 4 areas and overall quality of life perception and health status. The higher the total score is, the better quality of life is.
Stress level for overall health status self-evaluation | 6 weeks
  Stress level Questionnaire: Perceived Stress Scale, PSS-10. PPS-10 is rated on a 5-point likert scale where 0=Never, 1=Almost Never, 2=Sometimes, 3=Fairly Often, 4=Very Often. The higher the total score is, the more severe the stress level is.
Fatigue level for overall health status self-evaluation | 6 weeks
  Fatigue level Questionnaire: Fatigue Assessment Scale, FAS. FAS is a 10-item general fatigue questionnaire to assess fatigue. Five questions reflect physical fatigue and 5 questions (questions 3 and 6-9) mental fatigue.The total score of FAS ranges from 10 to 50. A total FAS score < 22 indicates no fatigue, a score ≥ 22 indicates fatigue.

CONTACTS AND LOCATIONS:
Overall Officials: Guoping YIN, Principal Investigator — Beijing Tsinghua Changgeng Hospital
Locations (1):
- Beijing Tsinghua Changgeng Hospital, Beijing, China